CLINICAL TRIAL: NCT06057402
Title: ELRANATAMAB POST TRIAL ACCESS: AN OPEN-LABEL, SINGLE-ARM STUDY FOR PARTICIPANTS WITH MULTIPLE MYELOMA CONTINUING FROM PFIZER-SPONSORED ELRANATAMAB CLINICAL STUDIES
Brief Title: Elranatamab Post Trial Access Study for Participants With Multiple Myeloma (MM)
Acronym: MagnetisMM15
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C1071015; 2023-505200-33-00 (Registry Identifier: CTIS (EU))
Record Dates: First submitted 2023-09-05; First posted 2023-09-28 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Multiple Myeloma
Keywords: Multiple Myeloma; Elranatamab; Post Trial Access; Roll-over Study; Extension Study; MM-15; MagnetisMM15; BCMA; BCMA antibody; Magnetism; Bispecific antibody; Elrexfio
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Elranatamab (Experimental): Elranatamab is a heterodimeric humanized full length bispecific IgG2 kappa antibody that targets BCMA on MM cells and CD3 on T cells
  Interventions: Drug: Elranatamab

INTERVENTIONS:
Drug: Elranatamab — Elranatamab is a heterodimeric humanized full-length bispecific IgG2 kappa antibody that targets BCMA on MM cells and CD3 on T cells
  Other Names: Elrexfio

SUMMARY:
This is a post-trial access (PTA) open-label, single-arm study in Multiple Myeloma participants who continue to derive clinical benefit from elranatamab monotherapy in the Pfizer-sponsored elranatamab Parent Studies.

DETAILED DESCRIPTION:
This is a single-arm elranatamab post-trial access study. Participants will receive elranatamab. All participants will receive elranatamab until disease progression, unacceptable toxicity, withdrawal of consent, study termination or, elranatamab becomes commercially accessible in the participant's country.

ELIGIBILITY:
Inclusion Criteria:

* Participants must agree to follow the reproductive criteria as outlined in the protocol
* Participants have completed a qualifying Parent Study, were still receiving elranatamab when the Parent Study terminated or completed, and are deriving clinical benefit from elranatamab (as determined by the investigator).

Exclusion Criteria:

* Any medical or psychiatric condition including recent (within the past year) or active suicidal ideation/behavior or laboratory abnormality that may increase the risk of study participation or, in the investigator's judgment, make the participant inappropriate for the study.
* Participants not previously enrolled or who have discontinued study treatment in a Parent Study are ineligible for participation in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-10-03 (Actual); Primary Completion 2032-02-22 (Estimated); Study Completion 2032-02-22 (Estimated)

PRIMARY OUTCOMES:
Incidence of nonserious adverse events (AEs) leading to permanent discontinuation | A minimum of 90 days after the last dose of study drug
Incidence of serious adverse events (SAEs) | A minimum of 90 days after the last dose of study drug

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (25):
- United States (14):
  - UCHealth Poudre Valley Hospital, Fort Collins, Colorado
  - UCHealth Harmony, Fort Collins, Colorado
  - UCHealth Greeley Hospital, Greeley, Colorado
  - Longs Peak Hospital, Longmont, Colorado
  - UCHealth Longs Peak Medical Center, Longmont, Colorado
  - UCHealth - Medical Center of the Rockies, Loveland, Colorado
  - Sylvester Comprehensive Cancer Center - The Lennar Foundation Medical Center, Coral Gables, Florida
  - University of Miami Hospital and Clinics Deerfield Beach, Deerfield Beach, Florida
  - Sylvester Comprehensive Cancer Center, Miami, Florida
  - University of Miami Hospital and Clinics - Griffin Cancer Research Building, Miami, Florida
  - University of Miami Hospital and Clinics, Miami, Florida
  - University of Michigan, Ann Arbor, Michigan
  - Henry Ford Cancer - Detroit (Brigitte Harris Cancer Pavilion), Detroit, Michigan
  - St. David's South Austin Medical Center, Austin, Texas
- Canada (3):
  - Arthur J.E. Child Comprehensive Cancer Centre, Calgary, Alberta
  - Cross Cancer Institute, Edmonton, Alberta
  - McGill University Health Centre, Montreal, Quebec
- China (4):
  - Peking University Third Hospital, Beijing, Beijing Municipality
  - Sun Yat-sen University Cancer Center, Guangzhou, Guangdong
  - Shandong Provincial Hospital, Jinan, Shandong
  - The first Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang
- Japan (2):
  - Japanese Red Cross Medical Center, Shibuya-ku, Tokyo
  - University Hospital,Kyoto Prefectural University of Medicine, Kyoto
- Taiwan (2):
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C1071015